CLINICAL TRIAL: NCT04463108
Title: A Description of Routine Treatment Pathways in a Cohort of Patients With Major Depression and "Active Suicidal Ideation With Intent" in Italy: the Arianna Observational Study.
Brief Title: A Study to Describe Routine Treatment Pathways in Participants With Major Depression and Active Suicidal Ideation With Intent in Italy
Acronym: ARIANNA
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108760; 54135419MDD4002 (Other: Janssen-Cilag S.p.A., Italy)
Record Dates: First submitted 2020-07-03; First posted 2020-07-09 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Major; Suicidal Ideation
MeSH Terms: conditions — Depressive Disorder, Major; Suicidal Ideation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with MDD and Active Suicidal Ideation with Intent: Participants with Major Depressive Disorder (MDD) and active suicidal ideation with intent as defined/confirmed by Investigator will be enrolled and treated in accordance with routine clinical practice. The primary data source for this study will be the medical records of each participant.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No intervention will be administered as a part of this study. Both retrospective and prospective data will be collected. The retrospective data will be collected through medical chart review.

SUMMARY:
The purpose of the study is to describe the pharmacological and non-pharmacological treatment utilization pathways in Italian routine clinical practice of participants with Major Depressive Disorder (MDD) and active suicidal ideation with intent.

ELIGIBILITY:
Inclusion Criteria:

* Participant must meet Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-5) diagnostic criteria for single episode or recurrent Major Depressive Disorder (MDD), based upon clinical assessment
* In the physician's opinion the current depressive episode is moderate-to-severe in terms of severity.
* In the physician's opinion, acute psychiatric hospitalization is clinically warranted due to participant's current active suicidal ideation with intent
* Participant must be capable of discernment
* Participant must be able to read and write in the Italian language
* Participant must have signed the informed consent form (ICF) indicating that he/she understands the study purpose and is willing to participate in the study
* Participant is in the site's catchment area, as evaluated by the Investigator

Exclusion criteria:

* Participant currently (that is, at the time of enrolment and based upon clinical assessment) meets DSM-5 criteria for psychotic disorder, bipolar or related disorders, antisocial personality disorder, borderline personality disorder, intellectual disability, autism spectrum disorder, dementia
* Participant meets the DSM-5 severity criteria for moderate or severe substance or alcohol use disorder (except for nicotine or caffeine) within the 6 months before enrolment, based upon clinical assessment
* Participant has participated in or is currently enrolled in any clinical trial with experimental treatments within the current major depressive episode

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population consists of participants with confirmed Major Depressive Disorder (MDD) and active suicidal ideation with intent as per physician's opinion.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2021-11-08 (Actual)

PRIMARY OUTCOMES:
Type of Comprehensive Treatment for Major Depression Disorder (MDD) and Active Suicidal Ideation with Intent | Up to 90 days
  Type of comprehensive treatment for MDD and active suicidal ideation with intent (for example, psychopharmacotherapy; psychosocial treatment; somatic therapy) will be reported.
Number of Psychiatric Drugs | Up to 90 days
  Number of psychiatric drugs (that is, polypsychopharmacy versus monotherapy) will be reported.
Duration of Treatment | Up to 90 days
  Duration of treatment for MDD and suicidal ideation with intent will be evaluated.
Sequence of Treatments in Participants with MDD and Suicidal Ideation with Intent | Up to 90 days
  Treatment sequences for participants with MDD and suicidal ideation with intent (for exapmple, administration of first-line antidepressant) will be assessed.
Care Setting | Up to 90 days
  Care setting (that is, in-patient and out-patient) will be assessed.

SECONDARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) Total Score | Up to Day 104 (End of Visit)
  The MADRS is a clinician-rated scale designed to measure changes in depression severity due to antidepressant treatment.The MADRS consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms) for a total possible score of 60. Higher scores represent a more severe condition.
European Quality of Life (EuroQol) 5-Dimension 5-Level Questionnaire (EQ-5D-5L) scores | Up to Day 104 (End of Visit)
  The EQ-5D-5L is a generic measure of health status. The EQ-5D-5L is a 5-item questionnaire that assesses 5 domains including mobility, self-care, usual activities, pain/discomfort and anxiety/depression plus a visual analog scale rating "health today" with anchors ranging from 0 (worst imaginable health state) to 100 (best imaginable health state).
Percentage of participants with AEs and SAEs | Up to Day 104 (End of visit)
  An adverse event (AE) is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. A Serious (AE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Healthcare Resource Utilization | Up to day 104 (End of Visit)
  Health Care Resource Utilization (HCRU) will be measured through the number of hospitalization visits, visits to the emergency department, inpatient hospitalization, specialist outpatient visits, number of day care visits, laboratory tests, instrumental and other diagnostic tests related to MDD with active suicidal ideation with intent.

OTHER OUTCOMES:
Suicidal ideation and behavior as Assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) Score | Up to Day 104 (End of study)
  Suicidal ideation or behavior will be measured using C-SSRS score. C-SSRS is a clinician rated assessment of suicidal behavior and/ or intent. Scale consists of 28 items in 4 sections: suicide behavior, actual attempts, suicidal ideation, and intensity of ideation. Suicidal ideation consists of 5 yes/no items: wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods (not plan) without intention to act, active suicidal ideation with some intent to act without specific plan, active suicidal ideation with specific plan and intent. Worsening of suicidal ideation will be an increase in severity of suicidal ideation from baseline.
Beck Hopelessness Scale (BHS) Score | Up to Day 104 (End of visit)
  BHS is paper-based self-reported measure to assess one's level of negative expectations or pessimism regarding future. The scale consists of 20 true-false items that examine the respondent's attitude over past week by either endorsing a pessimistic statement or denying an optimistic statement; 9-items are keyed false and 11 are keyed true. Items fall within 3 domains: feelings about future; loss of motivation; future expectations. Each response is assigned a score of 0 or 1. Total BHS score is sum of item responses, with range from 0 to 20, with a higher score representing higher level of hopelessness. Total scores that range from 0 to 3 are (normal range), scores 4 to 8 (mild hopelessness, scores 9 to 14 (moderate hopelessness), scores <14 (severe hopelessness). Negative change in score indicates improvement.
Montgomery-Asberg Depression Rating Scale Suicide Ideation: item 10 (MADRS-SI) | Up to Day 104 (End of Visit)
  MADRS is clinician-rated scale designed to measure depression severity, and to detect changes due to antidepressant treatment. MADRS item 10, or MADRS-SI evaluates apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts; scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of symptoms), summed for a total possible score of 0 to 60. Higher scores represent more severe condition.
Involvement Evaluation Questionnaire (IEQ) | Up to Day 104 (End of Visit)
  The 31-item Involvement Evaluation Questionnaire measures caregiver burden. It has been validated for caregivers of individuals with schizophrenia, covers a broad domain of caregiving consequences and refers to burden experienced within the past 4 weeks. Mean scores are calculated for the total scale and sub-scales. Total scores can range from 29 to 145 with sub-scale domains ranging - tension, 9-45; supervision, 6-30; worrying, 6-30; and urging, 8-40. Lower total and subscale scores indicate less burden and higher scores greater level of caregiver burden.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.p.A., Italy Clinical Trial, Study Director — Janssen-Cilag S.p.A.
Locations (24):
- Italy (24):
  - ASST Spedali Civili Brescia, Brescia
  - Ospedale Santissima Trinità, Cagliari
  - Ospedale Sant'Antonio Abate, Cantù
  - Ospedale Vittorio Emanuele, Catania
  - Ospedale Parodi Delfino, Colleferro
  - Ospedali Riuniti Foggia, Foggia
  - Ospedale San Giovanni di Dio, Frattamaggiore
  - Azienda Ospedaliera Universitaria San Martino di Genova, Genova
  - Az. USL 12 di Viareggio Ospedale Versilia, Lido di Camaiore
  - H.U. Santa Lucía, Macerata
  - ASST Fatebenefratelli Sacco, Milan
  - Ospedale Ca Granda - Niguarda, Milan
  - Dipartimento di Salute Mentale, Modena
  - Ospedale S Francesco d Assisi, Oliveto Citra
  - Aou San Luigi Gonzaga, Orbassano
  - Centro Salute Mentale, Padua
  - AOU Policlinico P.Giaccone, Palermo
  - P.O. Putignano, Putignano
  - Ospedale Infermi Rimini, Rimini
  - Azienda Ospedaliera Sant Andrea, Roma
  - Ospedale G. Mazzini, Teramo
  - A.O.U. Città della Salute e della Scienza, Torino
  - Azienda Sanitaria Universitaria Integrata di Udine, Udine
  - Azienda Ulss 8 Berica- Ospedale Di Vicenza, Vicenza

REFERENCES:
- [Derived] Pompili M, Dell'Osso BM, Rosso G, Amore M, Bellomo A, Mautone A, Pilotto E, Ramacciotti S, Scardigli MI, Ascione G, Cipelli R, Sansone C, Simoni L, Adami M, Delmonte D; ARIANNA Study Group. Routine treatment pathways in a cohort of patients with major depression and suicidality in Italy: the ARIANNA observational study. Compr Psychiatry. 2023 Nov;127:152430. doi: 10.1016/j.comppsych.2023.152430. Epub 2023 Oct 13. PMID 37837942